CLINICAL TRIAL: NCT06215976
Title: The Nephroprotective Effect of Metformin With Cisplatin in Bladder Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samah Essam Saber Mahran, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CL (3164)
Record Dates: First submitted 2023-12-16; First posted 2024-01-22 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Muscle-Invasive Bladder Carcinoma
Keywords: Metformin; cisplatin; nephroprotective effect; nephrotoxicity; bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator): (39) patients taking metformin (500 mg twice daily) with cisplatin (70 mg/m2) and gemcitabine (1000 mg/m2) (GC) protocol
  Interventions: Drug: Metformin Hydrochloride 500 MG
- Control (No Intervention): (39) patients taking cisplatin (70 mg/m2) gemcitabine (1000 mg/m2) (GC) protocol without metformin

INTERVENTIONS:
Drug: Metformin Hydrochloride 500 MG — Metformin 500mg tablets twice daily
  Arms: Metformin

SUMMARY:
The goal of this clinical trial is to evaluate the protective effect of metformin on nephrotoxicity of cisplatin in patients with bladder cancer. The main questions it aims to answer are:

* To determine protective effect of metformin on structural and functional kidney injury caused by cisplatin in patients with bladder cancer.
* To evaluate the safety of combining cisplatin and metformin on patients with bladder cancer

ELIGIBILITY:
Inclusion Criteria:

1. Non-diabetic adults of age between 18 to 65.
2. Chemotherapy naïve patients diagnosed with bladder cancer.
3. Patients with stable renal function: eGFR is above 60 ml/min/1.73 m2

Exclusion Criteria:

1. Patients with history of lactic acidosis.
2. Patients taking any nephrotoxic medication other than cisplatin (e.g., frusemide, NSAIDs, aminoglycoside or vancomycin).
3. Unstable renal function (defined as an increase in serum creatinine of 0.3 mg/dL or greater suddenly in 48 hours according to the acute kidney injury network (AKIN) classification
4. Patients with heart failure, acute myocardial infarction or cardiogenic collapse (shock).
5. Severe infection and sepsis.

   * Any infection requiring hospitalization.
   * Any infection leading to a need for oxygen, intubation, vasopressors or fluids to support blood pressure.
6. Alcohol intake.
7. Respiratory failure.
8. Severe hepatic impairment (Child-Pugh class C).
9. Patients with metastasis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
serum creatinine (SCr) | 12 week
  to assess the nephroprotective effect of metformin against cisplatin induced nephrotoxicity.
Human Neutrophil gelatinase-associated lipocalin (NGAL) | 12 week
  to assess the nephroprotective effect of metformin against cisplatin induced nephrotoxicity
Cystatin C | 12 week
  to assess the nephroprotective effect of metformin against cisplatin induced nephrotoxicity
Estimated glomerular filtration rate (eGFR) | 12 week
  to assess the nephroprotective effect of metformin against cisplatin induced nephrotoxicity

SECONDARY OUTCOMES:
FBG | 12 week
  to assess the safety of using cisplatin-metformin combination in bladder cancer patients receiving cisplatin
HbA1C | 12 week
  to assess the safety of using cisplatin-metformin combination in bladder cancer patients
Body weight | 12 week
  to assess the safety of using cisplatin-metformin combination in bladder cancer patients (monitoring weight loss)
Body Mass Index | 12 week
  to assess the safety of using cisplatin-metformin combination in bladder cancer patients (monitoring weight loss)
Blood pH | 12 week
  to assess the safety of using cisplatin-metformin combination in bladder cancer patients (monitoring lactic acidosis if any)
Blood Lactate Level | 12 week
  to assess the safety of using cisplatin-metformin combination in bladder cancer patients (monitoring lactic acidosis if any)

CONTACTS AND LOCATIONS:
Overall Officials: Samar Farid, Study Chair — faculty of pharmacy Cairo University
Locations (1):
- faculty of pharmacy Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Mahran SE, Salem SE, Sabry NA, Farid SF. The nephroprotective effect of metformin with cisplatin in bladder cancer: randomized clinical trial. Int Urol Nephrol. 2025 Nov;57(11):3611-3624. doi: 10.1007/s11255-025-04505-2. Epub 2025 May 3. PMID 40319155